CLINICAL TRIAL: NCT03080675
Title: Trial of a Nutritional Blend to Prevent Cognitive Decline in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 16.13.NRC; 2016-A01006-45, RC31/16/8196 (Registry Identifier: ANSM)
Record Dates: First submitted 2016-10-18; First posted 2017-03-15 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Cognitive Decline
Keywords: Aging population
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Nutritional blend of ingrédients including vitamins and fish oil
  Interventions: Dietary Supplement: Nutrional blend of ingredients including vitamins and fish oil
- Control comparator: (Placebo Comparator): control product does not contain any of the active ingredients and is matched for carbohydrate content to the active intervention.
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Nutrional blend of ingredients including vitamins and fish oil
  Arms: Experimental
Dietary Supplement: Control
  Arms: Control comparator:

SUMMARY:
To demonstrate the beneficial effects of 1-year intervention with a nutritional blend of ingredients on blood levels of nutritional biomarkers known to be linked with cognitive decline in non-demented adults with subjective memory concerns aged 70+ years

DETAILED DESCRIPTION:
This multicenter trial will be a placebo-controlled, double-blind, randomized, 2 parallel groups study. The subjects will be randomly allocated to one of two treatment groups (placebo or nutrition product). The duration of the intervention is 1 year.

The total sample size at baseline is 364 subjects, consisting of non-demented adults with subjective memory concerns aged 70+ years.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 70 years
2. Spontaneous memory complaints
3. Adequate fluency in the local language to understand the inform consent form and complete any other study document
4. Sufficient vision and hearing to complete study protocol procedures based on medical judgement
5. Has a study partner that is willing to participate as a source of information and has at least weekly contact with the participant (contact can be in-person, via telephone or electronic communication)
6. Has general health status that will not interfere with the ability to complete the study
7. Willing and able to participate and to give written consent to comply with study procedures
8. Willing to be informed in case a new clinical pathology is discovered through clinical examinations

Exclusion Criteria:

1. Exhibiting a loss of independence in basic activities of daily living (ADL score < 4)
2. MMSE score < 24
3. Dementia as determined by DSM-V criteria
4. Suffering from diseases that are likely to be life-threatening in the short-term
5. History or presence of a severe disease (e.g., cardiovascular, hepatic, renal (e.g., End Stage Renal Disease), gastroenteral, respiratory, endocrine, neurologic, psychiatric, immunologic, or hematologic disease or other conditions) that could, in the opinion of the investigator, interfere with the subjects safety or ability to complete the trial
6. Food allergy
7. Taking omega-3 dietary supplements containing >200 mg DHA per day during the last 6 months
8. Receiving or having received in the past 3 months a physician prescribed vitamin B12, B3 or vitamin B-complex
9. Receiving Alzheimer's Disease medication (Galantamine, Memantine Donezepil and Rivastigmine)
10. Deprived of their liberty by administrative or judicial decision, or under guardianship or admitted to a healthcare or social institution (subjects in non-assisted living facilities could be recruited).
11. Having participated in another clinical study in the previous month or is currently participating in another study.

    Subjects meeting one or more of the following criteria below will not be included in the PET scan and MRI-scan subset groups:
12. Wearing a pace-maker or having metal in the body which is exclusionary for MRI
13. Claustrophobic

Subjects who will participate in the PET-scan and MRI-scan subset groups, will be excluded for a 1-year period of any future projects involving investigations using ionizing radiation.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 362 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
Changes at 1 year in levels of nutritional risk factors involved in cognitive decline with ageing relative to baseline | [Time Frame: 1 year] [Safety Issue: No]
  Plasma erythrocyte-omega 3 index
Changes at 1 year in levels of nutritional risk factors involved in cognitive in cognitive decline with ageing relative to baseline | [Time Frame: 1 year] [Safety Issue: No]
  Homocysteine levels

SECONDARY OUTCOMES:
Change in cognitive function determined by a composite Z-score from 4 neuropsychological tests (see description) at 0, 6 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  The composite score combines the scores of the following neuropsychological tests: FCSRT score as the sum of free recall (sum of the three learning tests) and of cued recall (sum of free recall and indexed recall), Orientation score (10 items) from MMSE, Number of symbols reported during 90 sec (Digit symbol Substitution test) and the Number of words reported during 2-minutes (Category naming test)
Changes in cognitive function assessed by the FCSRT (Free and Cued Selective Reminding Test) at 0, 6 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  FCSRT score as the sum of free recall (sum of the three learning tests) and of cued recall (sum of free recall and indexed recall)
Changes in cognitive function assessed by the Orientation score from the Mini Mental Scale Examination (MMSE) at 0, 6 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  Orientation score: Subcale of MMSE (see outcome 8); score from 0 to 10.
Changes in cognitive function assessed by the WAIS-IV coding test at 0, 6 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  Number of symbols reported during 90 seconds
Changes in cognitive function assessed by the Category Naming Test (CNT) at 0, 6 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  Number of words reported during 2 minutes
Cognitive function assessed by the (Mini Mental Scale Examination) MMSE total score at 6 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  Total score of the MMSE from 0 to 30. Any score greater than or equal to 24 points (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment.
Cognitive status changes assessed by the Trail Making Test parts A and B at 0, 6 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  Time in sec to complete Trail Making Test parts A and B
Cognitive status changes assessed by the Logical Memory subtest of the WMS-R Test at 0, 6 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  Number of correct story elements recalled
Cognitive status changes assessed by the Letter Fluency Test at 0, 6 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  Number of correct words reported in 2 minutes
Cognitive status changes assessed by the Stroop Color Word Test (SCWT) at 0, 6 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  Time required to complete each sub-test and interference measure
Cognitive status changes assessed by the Digit Span (DS) at 0, 6 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  Number of digits recalled for forwards and backward sequences
Change in cognitive impairment assessed by the Clinical Dementia Rating - Sum of Boxes (CDR-SOB) at 0 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  CDR-SOB score ranging from 0 to 18 (0: Normal ; 0.5-4: Questionable cognitive impairment ; 4.5-9: Mild dementia ; 9.5-15.5: Moderate dementia ; 16-18: Severe dementia)
Change in clinical status assessed by Clinical Dementia Rating (CDR) at 0 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  Conversion rates to Mild cognitive impairment (MCI) and to dementia (0 = Normal, 0.5= very mild dementia, 1= mild dementia, 2 = moderate dementia, 3= severe dementia)
Subjective change in cognitive function assessed by the PROMIS Applied Cognition - Abilities instrument, Cognitive Function Instrument at 0, 1 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  PROMIS score: 33 items noted from 0 to 5 (Min score= 0, Max score =165) not used as diagnosis score but to assess the performance from baseline
Subjective change in quality of life and health status assessed by the EQ-5D-5L questionnaire at 0 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  EQ-5D-5L score: EQ-5D-5L, 5 item questionnaire and a visual analogue scale ranging from 0-100 to describe health status
Changes in depression status assessed by the Geriatric depression scale (GDS) at 0 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  GDS score ranging from 0 to 15: 0-9: Normal ; 10-19: Mild depression ; 20-30 : Severe depression.
Changes in depression, anxiety and psychiatric symptoms assessed by the Neuropsychiatric Inventory Questionnaire (NPI-Q) at 0 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  Change in the presence (yes-no) and severity score (1: mild; 2: moderate; 3: severe) of 12 neuropsychiatric symptoms related to dementia, as well as informant distress score for each of the present symptoms (from 0: 'No distress' to 5: 'Extreme distress') measured at 0 and 12 months.
Changes in physical functions assessed by the Short Physical Performance Battery (SPPB) at 0, 6 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  SPPB score ranging from 0 to 12. Assessment of score's evolution from baseline to 12 months.
Changes in frailty syndromes assessed by the Fried Frailty Criteria at 0 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  Grip strength, timed walking, involuntary weight loss, fatigue and physical activity (categories: robust, pre-frail, frail)
Changes in brain structure assessed by Magnetic Resonance Imaging (MRI) in a subset of the study population at 0 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  Regional tissue volume, Regional tissue thickness, Regional surface area, Intracranial volume (total, regional), Total brain volume, Regional volume (eg hippocampus)
Changes in brain structure assessed by fluid-attenuated inversion recovery (FLAIR) MRI and diffusion tensor imaging (DTI) in a subset of the study population at 0 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  Total white matter lesion volume
Changes in brain function assessed by Arterial spin label (ASL) perfusion MRI in a subset of the study population at 0 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  Cerebral blood flow
Changes in brain function assessed by resting State fMRI in a subset of the study population at 0 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  Brain connectivity
Changes in brain structure assessed by MRI diffusion tensor imaging (DTI) in a subset of the study population at 0 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  White matter integrity
Changes in brain function assessed by Amyloid Florbetapir Positron Emission Tomography (PET) in a subset of the study population at baseline | [Time Frame: 1 years] [Safety Issue: No]
  Amyloid load
Changes in levels of biomarkers associated with cognitive decline: BDNF levels at 0, 6 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  Brain-Derived Neurotrophic Factor (BDNF) plasma levels
Changes in levels of biomarkers associated with cognitive decline: Aβ40 levels at 0, 6 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  Aβ40 plasma levels
Changes in levels of biomarkers associated with cognitive decline: Aβ42 levels at 0, 6 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  Aβ42 plasma levels
Changes in levels of biomarkers associated with cognitive decline: Tau protein levels at 0, 6 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  Tau protein plasma levels
Changes in levels of biomarkers associated with cognitive decline: Asymmetric dimethylarginine levels at 0, 6 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  Asymmetric dimethylarginine plasma levels
Changes in levels of biomarkers associated with cognitive decline: Homocysteine levels at 0, 6 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  Homocysteine plasma levels
Changes in levels of blood plasma inflammatory markers 0, 6 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  Inflammatory markers (sCAMs, E-Selectin, TNF-alpha, IL1, IL6, IL10, CRP, neopterin)
Changes in levels of blood plasma markers of oxidative stress at 0, 6 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  Markers of oxidative stress (Oxidized Low-density lipoprotein (oxLDL), F2-isoprostane)
Changes in levels of plasma nutrient levels at 0, 6 and 12 months | [Time Frame: 1 year] [Safety Issue: No]
  e.g.vitamins, minerals, lipids, amino acids, erythrocyte omega-3 index
Treatment effects in a subgroup population defined by the below described subject characteristic: | [Time Frame: 1 year] [Safety Issue: No]
  Clinical Dementia Rating (CDR) of 0.5 at baseline
Treatment effects in a subgroup population defined by the below described subject characteristic: | [Time Frame: 1 year] [Safety Issue: No]
  Low DHA status (erythrocyte omega 3 index in the lower quartile) at baseline
Treatment effects in a subgroup population defined by the below described subject characteristic: | [Time Frame: 1 year] [Safety Issue: No]
  High plasma homocysteine levels (plasma homocysteine ≥ 12 µmol/L) at baseline
Treatment effects in a subgroup population defined by the below described subject characteristic: | [Time Frame: 1 year] [Safety Issue: No]
  CAIDE (Cardiovascular Risk Factors, Aging and Dementia) risk score at baseline
Treatment effects in a subgroup population defined by the below described subject characteristic: | [Time Frame: 1 year] [Safety Issue: No]
  Genotype

CONTACTS AND LOCATIONS:
Overall Officials: Bruno VELLAS, Principal Investigator — CHU Toulouse, Gérontopôle, Cité de la Santé, 20 Rue du Pont Saint Pierre, 31059 TOULOUSE Cedex 9
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No